CLINICAL TRIAL: NCT01621958
Title: Motor Training for Fall Prevention: Adaptation and Retention in Older Adults
Brief Title: Motor Training for Fall Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2001-0821; 5R01AG029616-03 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Fall Prevention
Keywords: balance loss; dynamic stability; motor learning; plasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor training (Experimental)
  Interventions: Behavioral: Repeated perturbation training
- Intensity control (Placebo Comparator)
  Interventions: Behavioral: Minimal perturbation training

INTERVENTIONS:
Behavioral: Repeated perturbation training — One session consisting of 24 slips total interspersed with 16 nonslip trials (1 block of 8 slips, 3 non-slips, 2nd block of 8 slips, 3 non-slips, a mixed block consisting of 8 slips and 10 non-slips). Retest consisting of one slip exposure at either 6 months, 9 months or 12 months.
  Other Names: Repeated slip training
  Arms: Motor training
Behavioral: Minimal perturbation training — One session consisting of a single slip exposure. Retest consisting of one slip exposure at either 6 months, 9 months or 12 months.
  Other Names: Single slip exposure
  Arms: Intensity control

SUMMARY:
Slip-related falls often cause injury; these often have catastrophic consequences, even among the healthiest older persons. Establishing a retainable preventive training regimen against slip-related falls would, without doubt, have major public health implications. In this study, investigators will demonstrate that older adults can significantly reduce their near-term risk of backward balance loss and falls through motor training with multiple protected slip exposure, and such adaptive improvements from such prophylactic training regimen can be retained over the course of a year.

DETAILED DESCRIPTION:
Slip-related falls often cause catastrophic injury for both frail and healthy older persons. Investigators have shown that, with motor training by repeated exposure to slips during walking, young adults are able to traverse a potential slipping hazard without losing their balance, regardless of whether a slip actually occurs or not. It is highly unlikely that these effects could be attributed to education or heightened awareness of the slipping threat alone. Furthermore, investigators have demonstrated that these improved motor skills acquired from a single session can be retained 4-6 months or longer upon re-testing, making such intervention highly attractive. Of greater interest, however, is the extent to which older adults can acquire and retain similar protective skills upon such training. This has not been tested to date. Also unknown is how potential confounding factors such as an older adult's functional status might interact with the training. These issues are of importance in that establishing a retainable preventive training regimen against slip-related falls would, without doubt, have major public health implications.

In this study, investigators will demonstrate that older adults can significantly reduce their near-term risk of backward balance loss and falls through motor training by repeated exposure to simulated slips interspersed with no-slip trials. Investigators will verify that awareness or observational learning alone cannot substitute for motor training through an awareness-control group. Investigators will then determine the extent to which adaptive improvements are retained over the course of a year. Finally, investigators will verify that although a single slip exposure may yield some retainable effect, this intensity control group will exhibit significantly less favorable long-term effect on the control of center of mass stability, body weight support, balance loss and fall upon slipping than the motor training group with repeated slips. In addition, investigator expect that the intensity-control group will also have a higher self-reported incidence of falls during the 12-month period than the motor training group with multiple slip exposure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no known history of musculoskeletal, neurological, cardiovascular, or pulmonary impairment that may affect their ability to perform the testing procedures will be included.
* Subjects in the balance-impaired group will specifically include subjects with unilateral or bilateral vestibular disorders and individuals with balance deterioration due to aging.
* Subjects in this group must be able ambulate independently for at least 5 meters and score 48/56 on the Berg Balance Scale, and must have no Central Nervous System disorders beyond vestibular disorders and no central/peripheral motor impairments.

Exclusion Criteria:

The exclusion criteria include the following:

1. using any sedative of any type,
2. having known history of osteoporosis,
3. having any clinically significant functional impairment related to a specific musculoskeletal, neurological, or cardiopulmonary disease,
4. ultrasound calcaneus bone mineral density T score < -1 (osteoporosis )
5. Mini-Mental State exam score < 25 (impaired cognition),
6. timed up-and-go > 13.5 sec (impaired mobility).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 212 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Fall incidence | 6 months

SECONDARY OUTCOMES:
Dynamic stability | 6 months
  The dynamic stability will be evaluated based on the dynamic relationship of motion state (i.e., the combination of position and velocity) between the center of mass and the base of support. It will be calculated as the shortest distance from the instantaneous motion state of the center of mass to the threshold against backward fall. It is a dimensionless variable.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chung Pai, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Clinical Gait and Movement Analysis Laboratory, Chicago, Illinois, United States